CLINICAL TRIAL: NCT01915199
Title: Effects of a Comprehensive Intervention on Blood Pressure Control in a Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: City of Turku (Other Government); Social Insurance Institution, Finland (Other)
Responsible Party: Principal Investigator, Teemu Niiranen, Medical Specialist, Finnish Institute for Health and Welfare
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVEL
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Critical Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients in this arm received a comprehensive intervention on hypertension through optimization of drug therapy, introduction of home blood pressure monitoring, and lifestyle guidance.
  Interventions: Other: Intensive Care
- Control (No Intervention): Patients randomized in this group did not receive any intervention and treatment continued according to conventional practice.

INTERVENTIONS:
Other: Intensive Care — Comprehensive intervention on hypertension through optimization of drug therapy, introduction of home blood pressure monitoring, and lifestyle guidance
  Arms: Intervention

SUMMARY:
The implementation of lifestyle modifications, home blood pressure (BP) measurement, and optimization of antihypertensive drug therapy have been shown to improve BP control in tightly controlled research settings. The investigators objective is to determine the effect of these interventions in a primary care setting, with the family practitioners and nurses serving as the interventionists. The investigaotrs hypothesis is that a comprehensive intervention performed in a primary care setting would lead to better blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-74 years
* Untreated office blood pressure of ≥ 160/100 mmHg or on active antihypertensive treatment.

Exclusion Criteria:

* Severe psychiatric or neurologic illnesses
* Heart failure (ejection fraction < 40% or previous hospitalization for heart failure)
* Hemodynamically significant valvular disease
* Unstable coronary heart disease
* Chronic kidney disease (proteinuria > 1 g/l or a serum creatinine concentration > 160 mmol/l)

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2000-10; Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Change in Office Systolic and Diastolic Blood Pressure | Baseline and at 12 Months.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Jula, MD, Principal Investigator — Finnish Institute for Health and Welfare; Teemu Niiranen, MD — Finnish Institute for Health and Welfare
Locations (1):
- Population Studies Unit, Turku, Finland

REFERENCES:
- [Result] Niiranen TJ, Leino K, Puukka P, Kantola I, Karanko H, Jula AM. Lack of impact of a comprehensive intervention on hypertension in the primary care setting. Am J Hypertens. 2014 Mar;27(3):489-96. doi: 10.1093/ajh/hpt204. Epub 2013 Nov 1. PMID 24186848